CLINICAL TRIAL: NCT02115815
Title: A Phase 1a Study to Evaluate the Safety of the Respiratory Syncytial Virus Vaccine MEDI7510 in Older Adults
Brief Title: A Study to Evaluate the Safety of the Respiratory Syncytial Virus Vaccine MEDI7510 in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CD-VA-MEDI7510-1134; BB-IND 15947 (Other: US FDA)
Record Dates: First submitted 2014-04-03; First posted 2014-04-16 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Respiratory Syncytial Virus (RSV); MEDI7510

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Placebo (Placebo Comparator): Sterile saline for human use from commercial source, liquid
  Interventions: Biological: Placebo
- RSV sF 20 mcg (Experimental): Participants will receive single dose of 20 mcg RSV sF by intramuscular injection on Day 1.
  Interventions: Biological: RSV sF 20 mcg
- MEDI7510 (20 mcg RSV sF) (Experimental): Participants will receive single dose of MEDI7510 (20 mcg RSV sF with 2.5 mcg glucopyranosyl lipid A [GLA] + 2% weight per volume stable emulsion) by intramuscular injection on Day 1.
  Interventions: Biological: MEDI7510 (20 mcg RSV sF)
- RSV sF 50 mcg (Experimental): Participants will receive single dose of 50 mcg RSV sF by intramuscular injection on Day 1.
  Interventions: Biological: RSV sF 50 mcg
- MEDI7510 (50 mcg RSV sF) (Experimental): Participants will receive single dose of MEDI7510 (50 mcg RSV sF with 2.5 mcg GLA + 2% weight per volume stable emulsion) by intramuscular injection on Day 1.
  Interventions: Biological: MEDI7510 (50 mcg RSV sF)
- RSV sF 80 mcg (Experimental): Participants will receive single dose of 80 mcg RSV sF by intramuscular injection on Day 1.
  Interventions: Biological: RSV sF 80 mcg
- MEDI7510 (80 mcg RSV sF) (Experimental): Participants will receive a single dose of MEDI7510 (80 mcg RSV sF with 2.5 mcg GLA + 2% weight per volume stable emulsion) by intramuscular injection on Day 1.
  Interventions: Biological: MEDI7510 (80 mcg RSV sF)

INTERVENTIONS:
Biological: Placebo — Participants will receive placebo (sterile saline for human use from commercial source liquid) on Day 1.
  Arms: Placebo
Biological: RSV sF 20 mcg — Participants will receive single dose of 20 mcg RSV sF by intramuscular injection on Day 1.
  Arms: RSV sF 20 mcg
Biological: MEDI7510 (20 mcg RSV sF) — Participants will receive single dose of MEDI7510 containing 20 mcg RSV sF by intramuscular injection on Day 1.
  Arms: MEDI7510 (20 mcg RSV sF)
Biological: RSV sF 50 mcg — Participants will receive single dose of 50 mcg RSV sF by intramuscular injection on Day 1.
  Arms: RSV sF 50 mcg
Biological: MEDI7510 (50 mcg RSV sF) — Participants will receive single dose of MEDI7510 containing 50 mcg RSV sF by intramuscular injection on Day 1.
  Arms: MEDI7510 (50 mcg RSV sF)
Biological: RSV sF 80 mcg — Participants will receive single dose of 80 mcg RSV sF by intramuscular injection on Day 1.
  Arms: RSV sF 80 mcg
Biological: MEDI7510 (80 mcg RSV sF) — Participants will receive single dose of MEDI7510 containing 80 mcg RSV sF by intramuscular injection on Day 1.
  Arms: MEDI7510 (80 mcg RSV sF)

SUMMARY:
The purpose of this study is to determine if the administration of single ascending intramuscular doses of the RSV sF antigen or MEDI7510 will be safe and well tolerated in adults 60 years or older who are healthy or who have stable, chronic underlying medical conditions.

DETAILED DESCRIPTION:
A phase 1a, first time in human, double-blind, randomized, placebo-controlled, cohort escalation study evaluating the safety and tolerability of a single ascending intramuscular dose of RSV sF or MEDI7510 or placebo.

Approximately 146 participants will be enrolled at 3 US study centers and randomized in a 5:1 ratio by cohort as described below:

Cohort 1: RSV sF 20 microgram (mcg) (n=20) or placebo (n=4) Cohort 1a: MEDI7510 (20 mcg RSV sF with 2.5 mcg glucopyranosyl lipid A (GLA) + 2% weight per volume stable emulsion (n=20) or placebo (n=4) Cohort 2: RSV sF 50 mcg (n=20) or placebo (n=4) Cohort 2a: MEDI7510 (50 mcg RSV sF with 2.5 mcg glucopyranosyl lipid A (GLA) + 2% weight per volume stable emulsion (n=20) or placebo (n=4) Cohort 3: 80 mcg RSV sF (n=20) or placebo (n=4) Cohort 3a: MEDI7510 (80 mcg RSV sF with 2.5 mcg glucopyranosyl lipid A (GLA) + 2% weight per volume stable emulsion (n=20) or placebo (n=4)

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 60 years
* Written informed consent and any locally required authorization obtained prior to any protocol related procedures
* Ambulatory or ambulatory with assistance (not institutionalized, bedridden, or homebound
* Weight at or above 110 Pounds (lbs)
* Hemoglobin within normal range for age and gender

Exclusion Criteria:

* History of allergy to any component of the vaccine
* Pregnancy or potential to become pregnant during the study. Females who have had a menstrual period within the 12 months prior to study enrollment or are undergoing any fertility treatment or who plan to undergo fertility treatments during the study period are excluded
* Any unstable chronic medical condition, including one that has resulted in change in therapy (medication or other) in the 30 days prior to randomization or hospitalization in the previous year or might be predicted to result in hospitalization in the year after enrollment. Participant with severe, untreated or uncontrolled underlying medical disease that might either compromise participant safety or affect the ability to assess safety of the investigational product are excluded
* Clinically significant abnormalities in Screening laboratory assessments or Screening electrocardiogram (ECG)
* History of hepatitis B or hepatitis C infection
* Cognitive disorder such that informed consent cannot be obtained directly from the participant
* Previous vaccination against respiratory syncytial virus (RSV)
* History of allergy to eggs in adulthood
* History of or current autoimmune disorder
* Immunosuppression caused by disease, including human immunodeficiency virus (HIV), or medications. Any oral prednisone dosing within 30 days of enrollment or planned dosing within the 360-day follow-up period would disqualify.
* History of splenectomy or of condition affecting splenic function
* History of cancer within preceding 5 years other than treated non-melanoma skin cancer
* Body Mass Index 40 or higher
* Significant infection or other acute illness, including fever over 100 fahrenheit (F) on the day prior to or day of randomization
* Receipt of any nonstudy vaccine within 30 days prior to study dosing or expected receipt of nonstudy vaccine within 30 days after study dosing
* Receipt of any investigational product in the 90 days prior to randomization or expected receipt of investigational product during the period of study follow-up
* Receipt of immunoglobulins or blood products within 4 months of study dosing (120 days) or expected receipt of investigational product during the period of study follow-up
* History of thrombocytopenia or bleeding disorder or use of anticoagulants. Participants receiving drugs with anti-platelet activity such as nonsteroidal antiinflammatory drugs, clopidogrel or aspirin are not excluded
* Expected receipt of antipyretic or analgesic medication on a daily or every other day basis from randomization through 72 hours after receipt of investigational product (IP) [a daily dose of 163 milligram (mg) or higher is not considered a contraindication to enrollment]
* Participants who have significant scarring, tattoos, abrasions, cuts, or infections over the deltoid region of both arms that, in the principle investigator's (PI) opinion, could interfere with evaluation of injection site local reactions
* Concurrent enrollment in another clinical study that involves any invasive clinical procedure, including phlebotomy
* History of alcohol or drug abuse or psychiatric disorder that in the PI's opinion would affect the participants safety or compliance with study
* Employees of individuals directly involved with the conduct of the study, individuals who themselves are involved with the conduct of the study, or immediate family members of such individuals.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Research Associates; Craig Curtis, MD, Principal Investigator — Compass Research; Steven Bart, MD, Principal Investigator — Accelovance; Judith Falloon, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Miami Research Associates, Miami, Florida
  - Compass Research, Orlando, Florida
  - Accelovance, Inc, Rockville, Maryland

REFERENCES:
- [Result] Falloon J, Ji F, Curtis C, Bart S, Sheldon E, Krieger D, Dubovsky F, Lambert S, Takas T, Villafana T, Esser MT. A phase 1a, first-in-human, randomized study of a respiratory syncytial virus F protein vaccine with and without a toll-like receptor-4 agonist and stable emulsion adjuvant. Vaccine. 2016 May 27;34(25):2847-54. doi: 10.1016/j.vaccine.2016.04.002. Epub 2016 Apr 19. PMID 27102821
- See also: CD-VA-MEDI7510-1134 Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2490&filename=MEDI7510-1134_Protocol_Legal%20IP_Redacted_04.05.16.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 246 subjects were screened. Of these, 146 subjects were enrolled.
Pre-assignment Details: A total of 146 participants were enrolled in the study. Of the 146 randomized participants, 2 participants did not receive investigational product. 144 participants were included in the As-treated Population.
Groups:
- Placebo: Participants received placebo (sterile saline for human use from commercial source, liquid) by intramuscular injection on Day 1.
- RSV sF 20 Microgram (mcg): Participants received single dose of 20 mcg RSV sF by intramuscular injection on Day 1.
- MEDI7510 20 Microgram (mcg): Participants received single dose of MEDI7510 (20 mcg RSV sF with 2.5 mcg glucopyranosyl lipid A [GLA] + 2% weight per volume stable emulsion) by intramuscular injection on Day 1.
- RSV sF 50 Microgram (mcg): Participants received single dose of 50 mcg RSV sF by intramuscular injection on Day 1.
- MEDI7510 50 Microgram (mcg): Participants received single dose of MEDI7510 (50 mcg RSV sF with 2.5 mcg GLA in 2% weight per volume stable emulsion) by intramuscular injection on Day 1.
- RSV sF 80 Microgram (mcg): Participants received single dose of 80 mcg RSV sF by intramuscular injection on Day 1.
- MEDI7510 80 Microgram (mcg): Participants received single dose of MEDI7510 (80 mcg RSV sF with 2.5 mcg GLA in 2% weight per volume stable emulsion) by intramuscular injection on Day 1.
Period: Overall Study
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Started | 24 | 20 | 20 | 20 | 20 | 22 | 20
Completed | 22 | 20 | 20 | 20 | 20 | 20 | 20
Not Completed | 2 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not enough drug to dose participant | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Missed appointment, randomized in error | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: As-treated Population (ATP): Participants who received any study investigational product were included in the ATP population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg) | Total
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 20 | 20 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.6 (7.6) | 66.5 (6.0) | 66.6 (4.1) | 69.3 (5.6) | 70.5 (6.1) | 70.0 (7.0) | 69.4 (7.0) | 68.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 9 | 10 | 10 | 8 | 11 | 68
  Male | 13 | 11 | 11 | 10 | 10 | 12 | 9 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Symptoms
Description: Solicited symptoms: tenderness or soreness at site of injection, pain at site of injection, fatigue or tiredness, headache, generalized muscle aches, swelling at the site of injection, redness at the site of injection, fever greater than or equal to (>=) 100.4 degrees F by any route from Day 1 to Day 7.
Time Frame: Day 1 to Day 7
Population: As-treated Population (ATP) included participants who received any study investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 20 | 20
participants | 6 | 4 | 15 | 7 | 14 | 9 | 17

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received investigational product. A serious adverse event (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of study product and Day 361 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From Day 1 to Day 28
Population: As-treated Population (ATP) included participants who received any study investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 20 | 20
participants
  TEAEs | 5 | 3 | 5 | 8 | 2 | 4 | 5
  TESAEs | 0 | 0 | 0 | 2 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events of Special Interest (TEAESIs), Treatment-Emergent Serious Adverse Events (TESAEs) and Treatment-Emergent New Onset Chronic Disease (NOCDs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received investigational product. A serious adverse event (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of study product and Day 361 that were absent before treatment or that worsened relative to pretreatment state. An AESI was one of scientific and medical interest specific to understanding of study product and may have required close monitoring and rapid communication by investigator to the sponsor. A NOCD was a newly diagnosed medical condition that is of a chronic, ongoing nature. It was observed after receiving investigational product and was assessed by investigator as medically significant.
Time Frame: From Day 1 to Day 361
Population: As-treated Population (ATP) included participants who received any study investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 20 | 20
participants
  TEAESIs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TESAEs | 2 | 0 | 0 | 5 | 1 | 3 | 0
  NOCDs | 2 | 0 | 0 | 4 | 1 | 4 | 2

4. Secondary Outcome: Post-dose Geometric Mean Titers (GMTs) From Baseline of Serum Antibodies Against Respiratory Syncytial Virus (RSV) by RSV A Microneutralization Assay
Description: RSV neutralizing antibody titers were measured using green fluorescent protein tagged RSV A 2
Time Frame: Baseline (Day 1), Day 29, 61, 91, 181, 271 and 361
Population: Immunogenicity population included participants in the As-treated population who had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and had baseline and/or any post-baseline result. Here, "n" is number of participants analysed for this outcome measure at give time points.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 20 | 20
titer
  Baseline (n= 24, 20, 20, 20, 20, 20, 20) | 441.37 [293.36 to 664.05] | 362.67 [252.96 to 519.95] | 367.73 [220.44 to 613.44] | 448.36 [282.62 to 711.28] | 442.03 [294.25 to 664.02] | 491.31 [327.84 to 736.30] | 428.16 [334.37 to 548.25]
  Day 29 (n= 24, 20, 20, 20, 19, 19, 20) | 430.04 [285.59 to 647.56] | 619.09 [419.12 to 914.45] | 809.84 [611.36 to 1072.77] | 981.61 [695.95 to 1384.51] | 1182.72 [813.02 to 1720.53] | 1116.48 [813.79 to 1531.74] | 1405.14 [1079.32 to 1829.32]
  Day 61 (n= 24, 20, 20, 20, 20, 20, 20) | 513.18 [339.82 to 775.00] | 716.09 [455.53 to 1125.70] | 764.04 [563.35 to 1036.21] | 959.74 [693.89 to 1327.44] | 1092.18 [769.39 to 1550.40] | 945.22 [732.16 to 1220.28] | 1046.60 [802.46 to 1365.04]
  Day 91 (n= 23, 20, 20, 19, 20, 19, 20) | 535.19 [350.79 to 816.54] | 635.83 [417.05 to 969.37] | 641.14 [464.88 to 884.24] | 849.22 [582.14 to 1238.85] | 1013.06 [700.41 to 1465.27] | 834.48 [626.96 to 1110.69] | 992.21 [799.35 to 1231.60]
  Day 181 (n= 23, 19, 20, 19, 20, 18, 20) | 373.79 [238.19 to 586.60] | 419.68 [281.38 to 625.97] | 421.09 [276.97 to 640.22] | 548.95 [372.94 to 808.01] | 487.07 [328.42 to 722.38] | 761.54 [558.06 to 1039.21] | 614.39 [435.55 to 866.66]
  Day 271 (n= 20, 20, 20, 19, 20, 17, 19) | 485.89 [325.78 to 724.69] | 600.28 [441.76 to 815.70] | 589.97 [418.92 to 830.86] | 829.32 [592.46 to 1160.89] | 710.41 [498.88 to 1011.61] | 705.14 [522.45 to 951.71] | 560.89 [360.47 to 872.76]
  Day 361 (n= 18, 0, 0, 0, 0, 17, 19) | 491.90 [313.90 to 770.85] | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | 675.04 [503.39 to 905.21] | 483.15 [360.07 to 648.30]

5. Secondary Outcome: Post-dose Geometric Mean Fold Rises (GMFRs) From Baseline of Serum Antibodies Against Respiratory Syncytial Virus (RSV) by RSV A Microneutralization Assay
Description: RSV neutralizing antibody titers were measured using green fluorescent protein tagged RSV A 2.
Time Frame: Day 29, 61, 91, 181, 271 and 361
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 20 | 20
fold rise
  Day 29 (n= 24, 20, 20, 20, 19, 19, 20) | 0.97 [0.89 to 1.07] | 1.71 [1.34 to 2.17] | 2.20 [1.43 to 3.39] | 2.19 [1.52 to 3.15] | 2.53 [1.85 to 3.46] | 2.51 [1.74 to 3.62] | 3.28 [2.51 to 4.29]
  Day 61 (n= 24, 20, 20, 20, 20, 20, 20) | 1.16 [0.95 to 1.42] | 1.97 [1.50 to 2.60] | 2.08 [1.33 to 3.25] | 2.14 [1.46 to 3.14] | 2.47 [1.74 to 3.51] | 1.92 [1.32 to 2.80] | 2.44 [1.88 to 3.18]
  Day 91 (n= 23, 20, 20, 19, 20, 19, 20) | 1.18 [0.99 to 1.39] | 1.75 [1.40 to 2.20] | 1.74 [1.14 to 2.67] | 2.01 [1.38 to 2.92] | 2.29 [1.65 to 3.18] | 1.72 [1.18 to 2.51] | 2.32 [1.82 to 2.95]
  Day 181 (n= 23, 19, 20, 19, 20, 18, 20) | 0.82 [0.72 to 0.94] | 1.13 [0.93 to 1.38] | 1.15 [0.69 to 1.90] | 1.30 [0.96 to 1.75] | 1.10 [0.89 to 1.37] | 1.50 [0.96 to 2.33] | 1.43 [1.10 to 1.87]
  Day 271 (n= 20, 20, 20, 19, 20, 17, 19) | 0.87 [0.76 to 0.99] | 1.66 [1.38 to 1.98] | 1.60 [1.02 to 2.53] | 1.96 [1.50 to 2.56] | 1.61 [1.29 to 2.00] | 1.38 [0.90 to 2.09] | 1.32 [0.89 to 1.95]
  Day 361 (n= 7, 0, 0, 0, 0, 17, 19) | 0.73 [0.58 to 0.91] | NA [NA to NA] — No participant was evaluated. | NA [NA to NA] — No participant was evaluated. | NA [NA to NA] — No participant was evaluated. | NA [NA to NA] — No participant was evaluated. | 1.32 [0.87 to 2.01] | 1.14 [0.91 to 1.42]

6. Secondary Outcome: Percentage of Participants Who Experience a Post-dose Seroresponse to Respiratory Syncytial Virus (RSV) by RSV A Microneutralization Assay
Description: Seroresponse defined as a greater than or equal to (>=) 4-fold rise from baseline.
Time Frame: Day 29
Population: Immunogenicity population included participants in the As-treated population who had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and had baseline and/or any post-baseline result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 19 | 19 | 20
percentage of participants | 0 [0.00 to 14.25] | 10.0 [1.23 to 31.70] | 5.0 [0.13 to 24.87] | 5.0 [0.13 to 24.87] | 10.5 [1.30 to 33.14] | 26.3 [9.15 to 51.20] | 25.0 [8.66 to 49.10]

7. Secondary Outcome: Post-dose Geometric Mean Titers (GMTs) From Baseline of Serum Antibodies Against Respiratory Syncytial Virus (RSV) by Anti-Fusion Protein (F) Immunoglobulin G (IgG) Assay
Description: Anti F IgG antibodies were determined by a multiplex IgG assay developed on the Meso Scale discovery platform.
Time Frame: Baseline (Day 1), Day 29, 61, 91, 181, 271 and 361
Population: Immunogenicity population included participants in ATP who had no protocol deviation judged to have potential to interfere with generation or interpretation of an immune response, and had baseline and/or any post-baseline result. Here, "n" is number of participants analysed for this outcome measure at give time points.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 20 | 20
titer
  Baseline (n= 24, 20, 20, 20, 20, 20, 20) | 64.89 [46.32 to 90.90] | 45.24 [30.89 to 66.26] | 64.94 [44.56 to 94.63] | 82.73 [44.45 to 153.97] | 93.51 [61.85 to 141.38] | 76.61 [45.39 to 129.29] | 73.84 [48.14 to 113.25]
  Day 29 (n= 24, 20, 20, 20, 20, 19, 20) | 66.16 [47.46 to 92.24] | 364.83 [214.31 to 621.05] | 658.97 [460.21 to 943.58] | 998.28 [636.44 to 1565.84] | 1159.03 [773.42 to 1736.89] | 924.44 [598.78 to 1427.22] | 1552.03 [1162.56 to 2071.99]
  Day 61 (n= 24, 20, 20, 20, 20, 20, 20) | 71.76 [53.17 to 96.85] | 351.98 [208.53 to 594.11] | 454.40 [316.95 to 651.45] | 738.48 [481.62 to 1132.34] | 875.86 [609.86 to 1257.88] | 731.83 [478.07 to 1120.28] | 1136.41 [834.01 to 1548.47]
  Day 91 (n= 22, 20, 20, 19, 20, 19, 20) | 71.57 [51.15 to 100.14] | 305.06 [184.64 to 504.02] | 365.38 [256.55 to 520.39] | 587.79 [376.03 to 918.81] | 704.64 [478.10 to 1038.52] | 596.80 [385.76 to 923.30] | 928.58 [675.84 to 1275.84]
  Day 181 (n= 23, 19, 20, 19, 20, 18, 20) | 68.41 [49.68 to 94.19] | 211.75 [134.85 to 332.50] | 235.81 [163.36 to 340.38] | 405.25 [252.75 to 649.78] | 456.76 [311.64 to 669.46] | 463.64 [311.06 to 691.06] | 604.90 [429.19 to 852.54]
  Day 271 (n= 20, 20, 20, 19, 20, 17, 19) | 78.65 [59.58 to 103.82] | 170.78 [116.92 to 249.46] | 196.53 [136.90 to 282.13] | 332.98 [209.95 to 528.11] | 358.67 [245.43 to 524.16] | 376.48 [256.43 to 552.75] | 364.40 [212.16 to 625.87]
  Day 361 (n= 18, 19, 20, 19, 20, 17, 19) | 73.17 [53.72 to 99.68] | 159.37 [110.50 to 229.87] | 186.26 [129.59 to 267.70] | 309.01 [196.87 to 485.03] | 298.08 [203.83 to 435.91] | 351.12 [245.76 to 501.67] | 374.98 [272.66 to 515.69]

8. Secondary Outcome: Post-dose Geometric Mean Fold Rises (GMFRs) From Baseline of Serum Antibodies Against Respiratory Syncytial Virus (RSV) by Anti-Fusion Protein (F) Immunoglobulin G (IgG) Assay
Description: Anti F IgG antibodies were determined by a multiplex IgG assay developed on the Meso Scale discovery platform.
Time Frame: Day 29, 61, 91, 181, 271 and 361
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 20 | 20
fold rise
  Day 29 (n= 24, 20, 20, 20, 20, 19, 20) | 1.02 [0.98 to 1.06] | 8.06 [4.51 to 14.41] | 10.15 [6.91 to 14.91] | 12.07 [6.29 to 23.14] | 12.39 [8.20 to 18.74] | 13.21 [7.59 to 22.99] | 21.02 [14.42 to 30.64]
  Day 61 (n= 24, 20, 20, 20, 20, 20, 20) | 1.11 [1.02 to 1.20] | 7.78 [4.40 to 13.75] | 7.00 [4.79 to 10.22] | 8.93 [4.63 to 17.22] | 9.37 [6.53 to 13.43] | 9.55 [5.48 to 16.67] | 15.39 [10.70 to 22.14]
  Day 91 (n= 22, 20, 20, 19, 20, 19, 20) | 1.11 [1.01 to 1.22] | 6.74 [3.96 to 11.47] | 5.63 [3.92 to 8.08] | 7.87 [4.16 to 14.89] | 7.54 [5.28 to 10.75] | 7.84 [4.43 to 13.86] | 12.58 [8.88 to 17.80]
  Day 181 (n= 23, 19, 20, 19, 20, 18, 20) | 1.08 [0.99 to 1.18] | 4.84 [3.11 to 7.55] | 3.63 [2.59 to 5.09] | 5.42 [2.86 to 10.29] | 4.88 [3.56 to 6.71] | 5.43 [3.12 to 9.43] | 8.19 [5.78 to 11.61]
  Day 271 (n= 20, 20, 20, 19, 20, 17, 19) | 1.04 [0.94 to 1.15] | 3.77 [2.54 to 5.60] | 3.03 [2.19 to 4.19] | 4.46 [2.48 to 8.02] | 3.84 [2.92 to 5.03] | 4.14 [2.40 to 7.12] | 5.12 [3.31 to 7.93]
  Day 361 (n= 18, 19, 20, 19, 20, 17, 19) | 1.05 [0.93 to 1.20] | 3.56 [2.42 to 5.23] | 2.87 [2.11 to 3.90] | 4.14 [2.40 to 7.14] | 3.19 [2.46 to 4.13] | 3.86 [2.27 to 6.57] | 5.27 [3.80 to 7.31]

9. Secondary Outcome: Percentage of Participants Who Experience a Post-dose Seroresponse to Respiratory Syncytial Virus (RSV) by Anti-Fusion Protein (F) Immunoglobulin G (IgG) Assay
Description: Seroresponse defined as a greater than or equal to (>=) 4-fold rise from baseline.
Time Frame: Day 29
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 19 | 20
percentage of participants | 0 [0.00 to 14.25] | 65.0 [40.78 to 84.61] | 90.0 [68.30 to 98.77] | 80.0 [56.34 to 94.27] | 90.0 [68.30 to 98.77] | 84.2 [60.42 to 96.62] | 100.0 [83.16 to 100.00]

10. Secondary Outcome: Post-dose Geometric Mean Counts (GMCs) From Baseline of T Cell Response Against Respiratory Syncytial Virus (RSV) by RSV F Enzyme-Linked Immunospot (ELISPOT)
Description: The ELISPOT assay for F protein-specific gamma interferon-producing T cells was performed using RSV F peptides.
Time Frame: Baseline (Day 1), Day 8 and 29
Population: Immunogenicity population included participants in ATP who had no protocol deviation judged to have potential to interfere with generation or interpretation of an immune response, and had baseline and/or any post-baseline result. Here, "N" and 'n' is number of participants analysed for this outcome measure and at given time points, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: spot forming counts per 10^6 PBMCs
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 24 | 20 | 20 | 20 | 20 | 19 | 20
spot forming counts per 10^6 PBMCs
  Baseline (n= 22, 16, 18, 19, 18, 20, 20) | 47.17 [38.28 to 58.14] | 41.59 [33.25 to 52.02] | 35.95 [31.13 to 41.52] | 39.81 [33.39 to 47.46] | 48.44 [38.90 to 60.31] | 37.78 [34.00 to 41.98] | 38.43 [33.51 to 44.07]
  Day 8 (n= 20, 20, 18, 17, 18, 15, 19) | 41.01 [34.29 to 49.05] | 62.63 [45.02 to 87.15] | 88.72 [53.16 to 148.06] | 80.25 [54.70 to 117.74] | 115.88 [66.23 to 202.76] | 88.59 [51.63 to 152.01] | 310.22 [179.10 to 537.34]
  Day 29 (n= 23, 16, 20, 19, 20, 19, 14) | 40.91 [32.90 to 50.88] | 39.93 [33.04 to 48.25] | 60.30 [42.19 to 86.19] | 69.36 [48.95 to 98.29] | 91.15 [60.37 to 137.62] | 77.13 [52.38 to 113.56] | 54.74 [33.43 to 89.64]

11. Secondary Outcome: Post-dose Geometric Mean Fold Rises (GMFRs) of T Cell Response Against Respiratory Syncytial Virus (RSV) by RSV F Enzyme-Linked Immunospot (ELISPOT)
Description: The ELISPOT assay for F protein-specific gamma interferon-producing T cells was performed using RSV F peptides.
Time Frame: Day 8 and 29
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 22 | 16 | 18 | 19 | 18 | 20 | 20
fold rise
  Day 8 (n= 20, 20, 18, 17, 18, 15, 19) | 0.90 [0.78 to 1.04] | 1.57 [1.10 to 2.24] | 2.18 [1.37 to 3.49] | 2.01 [1.29 to 3.12] | 2.21 [1.28 to 3.80] | 2.45 [1.46 to 4.10] | 8.01 [4.74 to 13.53]
  Day 29 (n= 23, 16, 20, 19, 20, 19, 14) | 0.88 [0.72 to 1.06] | 0.91 [0.77 to 1.07] | 1.54 [1.11 to 2.13] | 1.80 [1.25 to 2.58] | 1.99 [1.26 to 3.15] | 2.10 [1.47 to 2.99] | 1.36 [0.84 to 2.19]

12. Secondary Outcome: Percentage of Participants Who Experience a Post-dose 3-fold Cell-mediated Immune Response to RSV F on Day 8
Description: Seroresponse defined as a greater than or equal to (>=) 3-fold rise from baseline
Time Frame: Day 8
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Number analyzed (Participants) | 20 | 20 | 18 | 17 | 18 | 15 | 19
percentage of participants | 0 [0.00 to 17.65] | 12.5 [1.55 to 38.35] | 18.8 [4.05 to 45.65] | 25.0 [7.27 to 52.38] | 35.3 [14.21 to 61.67] | 46.7 [21.27 to 73.41] | 73.7 [48.80 to 90.85]

ADVERSE EVENTS:
Time Frame: AEs were collected from informed consent through Day 28 post dose; SAEs from informed consent through Days 28 and 361; treatment emergent adverse events of special interest and new onset chronic diseases through the Day 361 visit.
Arm/Group | Placebo | RSV sF 20 Microgram (mcg) | MEDI7510 20 Microgram (mcg) | RSV sF 50 Microgram (mcg) | MEDI7510 50 Microgram (mcg) | RSV sF 80 Microgram (mcg) | MEDI7510 80 Microgram (mcg)
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/20 | 0/20 | 5/20 | 1/20 | 3/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/24 | 3/20 | 5/20 | 8/20 | 2/20 | 4/20 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | RSV sF 20 Microgram (mcg) (N=20) | MEDI7510 20 Microgram (mcg) (N=20) | RSV sF 50 Microgram (mcg) (N=20) | MEDI7510 50 Microgram (mcg) (N=20) | RSV sF 80 Microgram (mcg) (N=20) | MEDI7510 80 Microgram (mcg) (N=20)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | RSV sF 20 Microgram (mcg) (N=20) | MEDI7510 20 Microgram (mcg) (N=20) | RSV sF 50 Microgram (mcg) (N=20) | MEDI7510 50 Microgram (mcg) (N=20) | RSV sF 80 Microgram (mcg) (N=20) | MEDI7510 80 Microgram (mcg) (N=20)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.